CLINICAL TRIAL: NCT01827774
Title: A Post-Market Study of Surgisis® Soft Tissue Graft for Repair of Pelvic Organ Prolapse
Brief Title: Soft Tissue Graft for Repair of Pelvic Organ Prolapse
Acronym: POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-015
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Graft repair
MeSH Terms: conditions — Pelvic Organ Prolapse

ARMS (1):
- Surgisis® Soft Tissue Graft (Experimental)
  Interventions: Device: Surgisis® Soft Tissue Graft

INTERVENTIONS:
Device: Surgisis® Soft Tissue Graft — Surgisis® Soft Tissue Graft for pelvic organ prolapse repair

SUMMARY:
The purpose of this Study is to collect information about the performance of the Surgisis® Soft Tissue Graft ("Study Product") for the repair of pelvic organ prolapse in women.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of transvaginal surgical repair of primary (i.e., de novo) pelvic organ prolapse.
* POPQ = stage 2 or 3 in the vaginal compartment with the leading edge of prolapse (i.e., more severe prolapse)
* At least one symptom associated with prolapse (e.g., any of the following including but not limited to vaginal bulge, vaginal pain/discomfort, voiding dysfunction, manual reduction (digitation) needed for defecation, fecal incontinence, dyspareunia)

Exclusion Criteria:

* Age < 18 years
* BMI > 40
* Not medically fit for transvaginal surgery under general or spinal anesthesia
* Active UTI at the time of the index procedure as determined by urine culture
* Vaginal atrophy (Note: Patient may be included after vaginal atrophy has been effectively treated.)
* Prior placement of synthetic mesh or biologic graft for pelvic organ prolapse
* A history of cervical, ovarian, uterine, endometrial, vaginal, vulval, colon, rectal or bladder cancer
* Currently planned obliterative surgical repair for pelvic organ prolapse
* Systemic infection at the time of surgery
* Requires chronic immunosuppressive therapy, including steroids or cytotoxic agents
* Pregnant, breastfeeding or planning pregnancy during the study period
* Previous diagnosis of collagen disorder (i.e., Marfan's, Ehlers-Danlos)
* Physical allergies or cultural objections to the receipt of porcine products
* Life expectancy of less than 12 months
* Ongoing participation in an investigational device or drug trial
* Currently undergoing evaluation or treatment for chronic pelvic pain (e.g., pain as a result of interstitial cystitis, endometriosis, vulvodynia, pelvic congestion syndrome)
* Active vaginal infection at the time of the index procedure
* History of pelvic inflammatory disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-03; Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

PRIMARY OUTCOMES:
Rate of recurrence of pelvic organ prolapse | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China